CLINICAL TRIAL: NCT01685697
Title: Comparison of Two Round Face Masks During Neonatal Resuscitation
Brief Title: Mask Ventilation With Different Face Masks During Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00033526
Record Dates: First submitted 2012-08-31; First posted 2012-09-14 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2017-01

CONDITIONS: Respiration; Insufficient or Poor, Newborn
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laerdal Mask (Active Comparator): Mask ventilation with a Laerdal face mask
  Interventions: Procedure: Mask ventilation with a Laerdal face mask
- F&P Mask (Experimental): Mask ventilation with a F&P face mask
  Interventions: Procedure: Mask ventilation with a F&P face mask

INTERVENTIONS:
Procedure: Mask ventilation with a Laerdal face mask — Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the intervention group.
  Arms: Laerdal Mask
Procedure: Mask ventilation with a F&P face mask — Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the control group.
  Arms: F&P Mask

SUMMARY:
Most premature babies have difficulty breathing at birth and need help (what we call resuscitation). The treatment for this is to gently inflate their lungs with a resuscitation device and a facemask. The device commonly used is a T-Piece infant resuscitator (which we call the T-Piece) and is used at The Royal Alexandra Hospital and all round the world.

To gentle inflate an infants lung the clinical team put a face mask around your baby's mouth and nose. The clinical team tries to achieve a good seal between the face and the mask. A problem of mask ventilation is that air can escape between the mask and the face (what we call mask leak). Currently, two different types of facemasks ("Laerdal mask" or "Fisher & Paykel mask") are routinely used in the delivery room at The Royal Alexandra Hospital.

The purpose of this study is to find out if one facemask is leaking less between the face and the mask.

DETAILED DESCRIPTION:
We will use a Laerdal round mask (Laerdal, Stavanger, Norway) compared to a Fisher & Paykel (FP) (Fisher & Paykel Healthcare, Auckland, New Zealand) 'round' neonatal resuscitation mask. The two point top hold for Laerdal 'round' mask and the rim hold for the Fisher & Paykel mask.

A Respiratory Function Monitor will be placed between the face mask and the ventilation device. It uses a small (dead space 1 mL) flow sensor to measure gas flow in and out of a face mask. This signal is automatically integrated to provide inspired and expired tidal volume. The difference equals the leak from the face mask. It also calculates respiratory rate and minute ventilation, measures spontaneous inspirations and ventilation pressures. The signals of airway flow, tidal volumes, airway pressure, inspired oxygen concentration, temperature, blood pressure, oxygen saturation, heart rate will be digitised and recorded at 200Hz using the Spectra physiological recording program (a customised neonatal respiratory physiology program).

We will compare the % of mask leak within the two face masks.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <32 weeks gestation born at The Royal Alexandra Hospital who require resuscitation in the delivery room will be recorded.

Exclusion Criteria:

* Infants will be excluded from final analysis if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation, including: Congenital Diaphragmatic Hernia. Infants will also be excluded if their parents refuse to give consent to this study.

Participants will be included in the first minutes after birth if they require mask ventilation for poor respiratory effort. Data will be collected from the Hospital chart until discharge at around 40 weeks gestation.

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD,PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Wood FE, Morley CJ, Dawson JA, Kamlin CO, Owen LS, Donath S, Davis PG. Improved techniques reduce face mask leak during simulated neonatal resuscitation: study 2. Arch Dis Child Fetal Neonatal Ed. 2008 May;93(3):F230-4. doi: 10.1136/adc.2007.117788. Epub 2007 Nov 26. PMID 18039750
- [Background] Chua C, Schmolzer GM, Davis PG. Airway manoeuvres to achieve upper airway patency during mask ventilation in newborn infants - An historical perspective. Resuscitation. 2012 Apr;83(4):411-6. doi: 10.1016/j.resuscitation.2011.11.007. Epub 2011 Nov 18. PMID 22101203
- [Background] Schmolzer GM, Morley CJ, Wong C, Dawson JA, Kamlin CO, Donath SM, Hooper SB, Davis PG. Respiratory function monitor guidance of mask ventilation in the delivery room: a feasibility study. J Pediatr. 2012 Mar;160(3):377-381.e2. doi: 10.1016/j.jpeds.2011.09.017. Epub 2011 Nov 5. PMID 22056350
- [Background] Schmolzer GM, Kamlin OC, O'Donnell CP, Dawson JA, Morley CJ, Davis PG. Assessment of tidal volume and gas leak during mask ventilation of preterm infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F393-7. doi: 10.1136/adc.2009.174003. Epub 2010 Jun 14. PMID 20547584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2013 to September 2013
Pre-assignment Details: The study used deferred consent approach. In this approach patient are randomized and asked to participant afterwards because of minimal risk to participation this study. Therefore there are a larger number of participant at the start date of the study and if they decline to participate a lower enrolled number.
Groups:
- Laerdal Mask: Mask ventilation with a Laerdal face mask
  Mask ventilation with a Laerdal face mask: Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the intervention group.
  Mask ventilation with a F&P face mask: Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the control group.
- F&P Mask: Mask ventilation with a F&P face mask
  Mask ventilation with a Laerdal face mask: Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the intervention group.
  Mask ventilation with a F&P face mask: Mask leak will be measured using a respiratory function monitor. Mask ventilation will be analyzed over a period of 5 minutes. The mean mask leak will be compared to the control group.
Period: Overall Study
Arm/Group | Laerdal Mask | F&P Mask
Started | 31 | 31
Completed | 28 | 28
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laerdal Mask | F&P Mask | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 28 | 56
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks]
  Gestational age in weeks | 28 (2) | 28 (3) | 28 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Leak
Description: Primary outcome: Difference in percentage of Leak
Time Frame: during mask ventilation in the first 5 minutes after birth
Measure: Median (Inter-Quartile Range); unit: % (percentage of mass leak)
Groups:
- Laerdal Mask; F&P Mask: Potentially eligible infants were randomized immediately prior to delivery and then received PPV as clinically necessary with either the F&P ∅35mm or ∅42mm F&P mask.
Arm/Group | Laerdal Mask | F&P Mask
Number analyzed (Participants) | 28 | 28
% (percentage of mass leak) | 35 [24 to 46] | 30 [25 to 36]

ADVERSE EVENTS:
Arm/Group | Laerdal Mask | F&P Mask
All-Cause Mortality (participants affected / at risk) | 2/28 | 2/28
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laerdal Mask (N=28) | F&P Mask (N=28)
Death during Admissions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No